CLINICAL TRIAL: NCT01364623
Title: An Open-label, Single and Multiple Application of Intranasal Testosterone Gel (TBS-2) in Healthy Premenopausal Female Subjects at Three Dose Levels
Brief Title: PK Study of Testosterone Nasal Gel (TBS-2) in Healthy Premenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBS-2-2011-01
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Female Sexual Dysfunction
Keywords: testosterone; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose TBS-2 single dose (Experimental): TBS-2 dispensers prefilled with 0.24% testosterone gel to deliver a single dose of 300 μg of testosterone per nostril, for a total dose of 600 μg given at 0800 hours (±30 minutes) on Day 2 of Period 1 for Cohort 1 (Low dose testosterone nasal gel, single dose)
  Interventions: Drug: Low dose testosterone nasal gel, single dose
- Medium dose TBS-2 single dose (Experimental): TBS-2 dispensers prefilled with 0.48% testosterone gel to deliver a single dose of 600 μg of testosterone per nostril, for a total dose of 1200 μg given at 0800 hours (±30 minutes) on Day 2 of Period 1 for Cohort 2 (Medium dose testosterone nasal gel, single dose)
  Interventions: Drug: Medium dose testosterone nasal gel, single dose
- High dose TBS-2 single dose (Experimental): TBS-2 dispensers prefilled with 0.72% testosterone gel to deliver a single dose of 900 μg of testosterone per nostril, for a total dose of 1800 μg given at 0800 hours (±30 minutes) on Day 2 of Period 1 for Cohort 3 (High dose testosterone nasal gel, single dose)
  Interventions: Drug: High dose testosterone nasal gel, single dose
- Medium dose TBS-2 multiple doses (Experimental): TBS-2 dispensers prefilled with 0.48% testosterone gel to deliver a single dose of 600 μg of testosterone per nostril, for a total dose of 1200 μg given t.i.d. daily at 0800 hours (± 30 minutes), 1600 hours (± 30 minutes), and 2400 hours (± 30 minutes) on Days 1 and 2 of Period 2, and once in the morning at 0800 hours (± 30 minutes) on Day 3 of Period 2 (Multi-dose group) (Medium dose testosterone nasal gel, multiple dose)
  Interventions: Drug: Medium dose testosterone nasal gel, multiple dose

INTERVENTIONS:
Drug: Low dose testosterone nasal gel, single dose — Low dose testosterone nasal gel, single dose
  Other Names: TBS-2
  Arms: Low dose TBS-2 single dose
Drug: Medium dose testosterone nasal gel, single dose — Medium dose testosterone nasal gel, single dose
  Other Names: TBS-2
  Arms: Medium dose TBS-2 single dose
Drug: High dose testosterone nasal gel, single dose — High dose testosterone nasal gel, single dose
  Other Names: TBS-2
  Arms: High dose TBS-2 single dose
Drug: Medium dose testosterone nasal gel, multiple dose — Medium dose testosterone nasal gel, multiple dose
  Other Names: TBS-2
  Arms: Medium dose TBS-2 multiple doses

SUMMARY:
The purpose of this study was to assess the bioavailability of total testosterone through pharmacokinetic profiles obtained following (a) single administration of three doses of TBS-2 b) multiple administration TBS-2.

In addition, assessing the bioavailability of free testosterone, dihydrotestosterone, SHBG and estradiol through pharmacokinetic profiles was also conducted.

DETAILED DESCRIPTION:
This is a 2 Period study that requires overnight stays in clinic. Blood samples are required at all visits including sampling at predefined time periods during the overnight stays.

Period I

Subjects were checked-in on Day 1 Period I to start their baseline testosterone measurement (dependant on menstrual cycle, preferably within 48hr of start of the menstrual cycle). They remained institutionalized until Day 4 morning, and were checked out after the 48 hour blood draw and study close-out for those that did not continue with Period II.

Period II (Multi-Dose)

At the end of Period 1, a total of 8 subjects sampled from these 3 cohorts, who were willing and able to continue with the multiple-dose portion of the study were selected to participate in Period 2. Subjects were institutionalized starting on Day 1 of Visit 3 until Day 5 morning of Visit 3, and were checked out after the 48 hour blood draw and study close-out.

ELIGIBILITY:
Inclusion Criteria

* Subjects having regular menstrual cycles between 26-32 days.
* Women of childbearing potential must agree to use one of the following reliable birth control methods prior to the study, during the study and up until one month after the end of the study:

  * Surgically sterile
  * Intrauterine device in place for at least 3 months prior to study initiation
  * Barrier method (condom with spermicidal agent use by partner)
  * Abstinence
* Negative for drugs of abuse, hepatitis B-surface antigen, hepatitis C, HIV, and pregnancy (serum ß-HCG).
* Body Mass Index greater than or equal to 18.5 kg/m² and less than or equal to 35 kg/m².
* Subjects with a normal ENT exam.
* Subjects with normal TSH values.
* No clinically significant findings in the physical examination, 12-lead ECG and vital signs
* Normal thyroid function. Physiological prolactin concentration.
* All clinical laboratory test values within the acceptable ranges (any clinically significant findings will require investigator/sponsor approval)
* Able to understand and provide written informed consent.
* Availability of the subject for the entire study period and willingness of the subject to adhere to protocol requirements, as evidenced by a signed ICF

Exclusion Criteria

* Known history of hypersensitivity to Testosterone (e.g. Intrinsa patch) and/or related drugs.
* Known history of polycystic ovarian syndrome.
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, psychiatric, hematological, reproductive, liver or kidney disease, unless judged not clinically significant by the Principal Investigator or medical designate.
* Presence of or known history of Estrogen-responsive tumors such as breast cancer and /or history of any cancer, excluding basal cell carcinoma.
* Known history of frequent clinically significant acne.
* Known history of hirsutism
* History of nasal surgery, specifically turbinoplasty, septoplasty, rhinoplasty, "nose job", or sinus surgery.
* Prior nasal fractures.
* Active allergies, such as rhinitis, rhinorrhea, and nasal congestion.
* Mucosal inflammatory disorders, specifically pemphigus, and Sjogren's syndrome.
* Sinus disease, specifically acute sinusitis, chronic sinusitis, or allergic fungal sinusitis.
* History of nasal disorders or sleep apnea.
* Use of any form of intra-nasal medication delivery, specifically nasal corticosteroids and oxymetazoline containing nasal sprays
* History of Hepatitis B, a positive test for Hepatitis B surface antigen, a history of Hepatitis C, a positive test for Hepatitis C antibody, a history of HIV infection or demonstration of HIV antibodies.
* Any history of severe allergic reaction (including drugs, food, insect bites, environmental allergens or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any history of drug abuse or alcohol abuse as per DSM-IV criteria within 6 months of study drug administration.
* Current treatment with any hormone replacement therapy within previous 12 months, treatment with drugs which interfere with metabolism of Testosterone within 30 days of study drug administration and/or any other prescription medications. Difficulty in abstaining from OTC medication for the duration of study.
* Use of oral, transdermal and implant contraceptives within 30 days prior to drug administration or a depot contraceptives injection within one year prior to drug administration.
* Evidence of pregnancy or lactation.
* Subjects who are breast feeding or have breast fed within the last six (6) months prior to the Screening Visit.
* Administration of another investigational drug within 30 days prior to study medication administration.
* Blood donation within 56 days prior to study medication administration.
* Any participation as a plasma donor in a plasmapheresis program within seven days preceding screening in this study.
* Intolerance to venipuncture.
* History of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation.
* History of Deep Venous Thrombosis or coagulation disorders.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Tkachenko, MD, Study Director — Trimel Pharmaceuticals Corporation
Locations (1):
- Premier Research International LLC, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose TBS-2 Single Dose: Low dose testosterone nasal gel: Single dose administration
- Medium Dose TBS-2 Single Dose: Medium dose testosterone nasal gel: Single dose administration
- High Dose TBS-2 Single Dose: High dose testosterone nasal gel: single dose administration
- Medium Dose TBS-2 Multiple-Dose: High dose testosterone nasal gel: multiple dose administration
Period: Single Dose
Arm/Group | Low Dose TBS-2 Single Dose | Medium Dose TBS-2 Single Dose | High Dose TBS-2 Single Dose | Medium Dose TBS-2 Multiple-Dose
Started | 8 | 8 | 8 | 0
Completed | 8 | 8 | 8 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Multiple Dose
Arm/Group | Low Dose TBS-2 Single Dose | Medium Dose TBS-2 Single Dose | High Dose TBS-2 Single Dose | Medium Dose TBS-2 Multiple-Dose
Started | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose TBS-2: Low dose testosterone nasal gel: Single dose administration
- Medium Dose TBS-2: Medium dose testosterone nasal gel: Single dose administration
  Medium dose testosterone nasal gel: Multiple dose administration
- High Dose TBS-2: High dose testosterone nasal gel: Single dose administration
- Total: Total of all reporting groups
Arm/Group | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (5.73) | 29.8 (4.43) | 27.0 (6.57) | 29.8 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 4 | 11
  Not Hispanic or Latino | 6 | 3 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 7 | 6 | 6 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bioavailability (AUC0-t) of Total Testosterone Through Pharmacokinetic (PK) Profiles
Description: Area under the concentration time curve from time zero to the last measurable concentration time point (AUC0-t) for single dose and AUCtau shown for multiple dose.
Time Frame: Based on blood samples collected -0.25, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 16, 20, 23.5h relative to dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/dL
Groups:
- Medium Dose TBS-2 Multiple-Dose: Medium dose testosterone nasal gel: Multiple dose administration
Arm/Group | Low Dose TBS-2 Single Dose | Medium Dose TBS-2 Single Dose | High Dose TBS-2 Single Dose | Medium Dose TBS-2 Multiple-Dose
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/dL | 223.981 (39) | 328.002 (35.8) | 834.391 (49.7) | 553.325 (41.4)

2. Primary Outcome: Bioavailability (Cmax) of Total Testosterone Through Pharmacokinetic Profiles
Description: Cmax - maximum concentration of total testosterone observed after dosing of TBS-2
Time Frame: Based on blood samples collected -0.25, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 16, 20, 23.5h relative to dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Groups:
- Low Dose TBS-2 - Single Dose: Low dose testosterone nasal gel: Single dose administration
- Medium Dose TBS-2 - Single Dose: Medium dose testosterone nasal gel: Single dose Administration
- High Dose TBS-2 - Single Dose: High dose testosterone nasal gel: single dose Administration
- Medium Dose TBS-2 - Multiple Dose: Medium dose testosterone nasal gel: multiple dose administration
Arm/Group | Low Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Single Dose | High Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/dL | 34.058 (61.1) | 62.880 (48.6) | 113.912 (44.3) | 137.555 (41.5)

3. Primary Outcome: Medium Dose TBS-2 Multiple Dose Average Steady-state Concentration (Cavg) of Total Testosterone
Time Frame: -0.25, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48h after Day 3 dosing
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Medium Dose TBS-2 - Multiple Dose: Medium dose testosterone nasal gel - multiple dose administration:
  A total dose of 1200 μg given t.i.d. daily at 0800 hours (± 30 minutes), 1600 hours (± 30 minutes), and 2400 hours (± 30 minutes) on Days 1 and 2 of Period 2, and once in the morning at 0800 hours (± 30 minutes) on Day 3 of Period 2).
Arm/Group | Medium Dose TBS-2 - Multiple Dose
Number analyzed (Participants) | 8
ng/dL | 0.944 (0.408)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) for Dihydrotestosterone Following TBS-2
Description: AUCt shown for single dose and AUCtau for multiple dose.
Time Frame: Based on blood samples collected -0.25, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 16, 20, 23.5h relative to dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/dL
Arm/Group | Low Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Single Dose | High Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/dL | 23.515 (74.9) | 38.457 (49.1) | 85.180 (64.2) | 122.194 (40.0)

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) for Estradiol Following TBS-2
Description: AUCt shown for single dose and AUCtau for multiple dose.
Time Frame: Based on blood samples collected -0.25, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 16, 20, 23.5h relative to dosing
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Low Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Single Dose | High Dose TBS-2 - Single Dose | Medium Dose TBS-2 - Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 8
pg*h/mL | 105.763 (118.7) | 75.97 (82.2) | 43.97 (197.9) | 400.264 (54.0)

ADVERSE EVENTS:
Time Frame: 36 days
Groups:
- Medium Dose TBS-2 Multiple Dose: Medium dose testosterone nasal gel: multiple dose administration
Arm/Group | Low Dose TBS-2 Single Dose | Medium Dose TBS-2 Single Dose | High Dose TBS-2 Single Dose | Medium Dose TBS-2 Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8 | 3/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose TBS-2 Single Dose (N=8) | Medium Dose TBS-2 Single Dose (N=8) | High Dose TBS-2 Single Dose (N=8) | Medium Dose TBS-2 Multiple Dose (N=8)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 1 | 1 | 0
Catheter site hemorrhage (General disorders) | 0 | 0 | 2 | 0
Catheter site inflammation (General disorders) | 2 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 1
Vulvitis (Infections and infestations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No